CLINICAL TRIAL: NCT00247611
Title: Changing ART Adherence Behavior: The Lifewindows Project
Brief Title: Improving Treatment Adherence in HIV-Infected Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Fisher, Principal Investigator, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH066684 (NIH); R01MH066684 (NIH); DAHBR 9A-ASPG
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-11

CONDITIONS: HIV Antiretroviral Therapy (ART) Adherence; Health Behavior
Keywords: HIV; AIDS; Antiretroviral Medication Adherence
MeSH Terms: conditions — Health Behavior; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): Participants will receive the control condition
  Interventions: Other: Control
- Intervention (Experimental): Participants will receive the LifeWindows Intervention sessions
  Interventions: Behavioral: LifeWindows Intervention Sessions

INTERVENTIONS:
Behavioral: LifeWindows Intervention Sessions — At each clinical care visit, intervention arm participants use the full LifeWindows program, which includes welcome and assessment surveys and also includes the active intervention modules. ART adherence promotion intervention activities are tailored to the participant's assessment responses. Participants select which activities he or she wishes to use which culminates in an adherence specific goal.
  Arms: Intervention
Other: Control — At each clinical care visit, control arm participants use the portion of the LifeWindows software program that provides a welcome from the avatar and collection of assessment items/surveys.
  Arms: Control

SUMMARY:
This study will develop and evaluate the efficacy of an individualized, interactive, computer software program delivered in conjunction with clinical care in increasing and supporting antiretroviral therapy adherence in HIV-infected individuals.

DETAILED DESCRIPTION:
When antiretroviral therapy (ART) is taken correctly, it can dramatically improve the health and well-being of HIV-infected individuals. However, when the treatment regimen is not followed carefully, the therapy can be ineffective in managing one's HIV, and also can allow for the development of strains of HIV that may be resistant to treatment. Effective ART adherence interventions can help patients to avoid potentially serious individual and public health consequences of suboptimal adherence, but such interventions are often expensive and too intensive for clinics to support offering over time to their patients. This study will develop and evaluate the effectiveness of an individualized, interactive, computer-software intervention program delivered in clinical care in increasing ART adherence in HIV-infected individuals. Because the intervention is a software program, clinic resources required for implementation and sustaining availability over time are minimized.

Participants in this ~18-month study were recruited from one of 5 participating clinics that provide HIV care and randomly assigned to control (an assessment only version of the software) or intervention (assessment and tailored intervention software) arm. Participants completed their assigned task in concert with their regularly scheduled HIV medical care visits (but no more frequently than once a month). Primary outcomes were measured at each medical visit. The effect of the adherence intervention was evaluated through comparison of treatment and control arm adherence reports over time and VL.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* English-speaking
* Currently receiving treatment at one of the participating sites
* Currently receiving antiretroviral therapy

Exclusion Criteria:

* Marked cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D. Fisher, PhD, Principal Investigator — University of Connecticut; K. Rivet Amico*, PhD, Principal Investigator — University of Connecticut (*co-PI); Deborah H. Cornman*, PhD, Principal Investigator — University of Connecticut (*co-PI); William A. Fisher*, PhD, Principal Investigator — University of Western Ontario (*co-PI)
Locations (5):
- United States (5):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Yale-New Haven Hospital Nathan Smith Clinic, New Haven, Connecticut
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Waterbury Hospital, Waterbury, Connecticut

REFERENCES:
- [Result] Fisher JD, Amico KR, Fisher WA, Cornman DH, Shuper PA, Trayling C, Redding C, Barta W, Lemieux AF, Altice FL, Dieckhaus K, Friedland G; LifeWindows Team. Computer-based intervention in HIV clinical care setting improves antiretroviral adherence: the LifeWindows Project. AIDS Behav. 2011 Nov;15(8):1635-46. doi: 10.1007/s10461-011-9926-x. PMID 21452051
- See also: PubMed record of results article — http://www.ncbi.nlm.nih.gov/pubmed/21452051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV + patients were recruited via provider referral and notices about the study posted in five large HIV care clinics in Connecticut, USA.
Period: Baselined
Arm/Group | Control | Intervention
Started | 304 (Participants randomized) | 290 (Participants randomized)
Completed | 287 (Randomized participants who completed at least 2 adherence assessments/sessions) | 277 (Randomized participants who completed at least 2 adherence assessments/sessions)
Not Completed | 17 | 13
Not completed — Completed baseline, never placed on ARVs | 8 | 5
Not completed — Completed baseline only | 9 | 8
Period: Intention to Treat Sample
Arm/Group | Control | Intervention
Started | 304 (Participants randomized) | 290 (Participants randomized)
Completed | 287 (Randomized participants who completed at least 2 adherence assessments/sessions) | 277 (Randomized participants who completed at least 2 adherence assessments/sessions)
Not Completed | 17 | 13
Period: On Protocol Sample
Arm/Group | Control | Intervention
Started | 287 (ITT sample participants) | 277 (ITT sample participants)
Completed | 176 (Participants with no interruptions in ART receipt and completing 6 or more LifeWindows assessments) | 152 (Participants with no interruptions in ART receipt and completing 6 or more LifeWindows assessments)
Not Completed | 111 | 125

BASELINE CHARACTERISTICS:
Population: Baseline characteristics provided for randomized sample. Analyses were conducted on those with >=2 adherence assessments for ITT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 304 | 290 | 594
Age, Categorical [Count of Participants; unit: Participants] — Intent to Treat (ITT) Sample
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 301 | 284 | 585
    >=65 years | 3 | 6 | 9
Age, Categorical [Number; unit: participants] — On Protocol (OP) The On-Protocol sample was derived from the ITT sample who also had completed >=6 assessments and had no ART receipt interruptions.
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 174 | 149 | 323
    >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Intent to Treat (ITT) Sample
  years | 47.28 (8.01) | 46.76 (8.00) | 47 (8)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent to Treat (ITT) Sample
  Participants
    Female | 119 | 110 | 229
    Male | 185 | 180 | 365
Gender [Number; unit: participants] — On Protocol (OP)
  participants
    Female | 72 | 66 | 138
    Male | 104 | 86 | 190
Region of Enrollment [Number; unit: participants] — Intent to Treat (ITT) Sample
  participants
    United States | 304 | 290 | 594

OUTCOME MEASURES:

1. Primary Outcome: AIDS Clinical Trials Group (ACTG) 3-day Recall Measure of Doses Taken
Description: This measure asks participants to report the number of doses taken on each of the past 3-days, relative to number he or she was prescribed to take, and produces a % adherence score. For this study, adherence over the past 3-days was established for each medication separately then averaged over the full regimen. For main outcomes, perfect vs imperfect adherence was evaluated. Significant findings on perfect/imperfect adherence were followed with sensitivity tests to determine if lowest threshold (eg., 90%, 80%, 70% adherence) effect was maintained.
  See: Chesney MA, Ickovics JR, Chambers DB, et al. Self-reported adherence to antiretroviral medications among participants in HIV clinical trials: the AACTG adherence instruments. Patient care committee & adherence working group of the outcomes committee of the adult AIDS clinical trials group (AACTG). AIDS Care. 2000;12(3):255-266.
Time Frame: Measured at each clinical care visit over 18 months of participation
Population: Intent to treat included all participants with >=2 adherence assessments; OP sample further restricted this sample to those with >=6 assessments and no treatment interruptions over 18-months of participation. Multiple pairwise comparison replaced missing values. HLM was used for over-time analyses on proportion reporting perfect adherence.
Measure: Number; unit: percent with 100% adherence
Groups:
- Control (ITT Sample %): 287 (94%) of the 304 randomized to control
- Intervention (ITT Sample): 277 (96%) of the 290 randomized to Intervention condition
- Control (On Protocol Sample): 176 (61%) of the ITT included control arm participants
- Intervention (On Protocol): 152 (55%) of the ITT included intervention arm participants
Arm/Group | Control (ITT Sample %) | Intervention (ITT Sample) | Control (On Protocol Sample) | Intervention (On Protocol)
Number analyzed (Participants) | 287 | 277 | 176 | 152
percent with 100% adherence
  1 LifeWindows Visit (%) | 72.89 | 75.46 | 74.86 | 77.33
  2 LifeWindows Visits (%) | 80.36 | 82.48 | 81.50 | 85.53
  3 LifeWindows Visits (%) | 81.15 | 80.16 | 84.09 | 84.11
  4 LifeWindows Visits (%) | 79.92 | 81.78 | 80.11 | 81.58
  5 LifeWindows Visits (%) | 83.41 | 87.13 | 82.86 | 88.74
  6 LifeWindows Visits (%) | 81.25 | 82.46 | 81.61 | 83.55
  7 LifeWindows Visits (%) | 79.73 | 85.61 | 79.70 | 87.18
  8 LifeWindows Visits (%) | 79.82 | 88.54 | 79.00 | 91.76
  9 LifeWindows Visits (%) | 82.02 | 87.14 | 81.58 | 89.39
  10 LifeWindows Visits (%) | 69.12 | 80.70 | 71.93 | 84.62
  11 LifeWindows Visits (%) | 70.21 | 78.57 | 68.42 | 83.78
  12 LifeWindows Visits (%) | 78.13 | 90.63 | 73.08 | 88.46
  13 LifeWindows Visits (%) | 68.00 | 87.50 | 65.00 | 85.71
  14 LifeWindows Visits (%) | 69.23 | 85.71 | 70.00 | 81.82
Statistical Analysis 1: Comparison: Control (ITT Sample %) vs Intervention (ITT Sample); For the ITT sample, the observed pattern of an increasing proportion of participants in the intervention arm reporting perfect adherence as time progressed from was associated with a p-value of 0.12, two-tailed alpha 0.05; Test type: Superiority or Other; p = 0.12, HLM — The p-value was not adjusted for multiple comparisons, and thresholds for significance were 0.05 alpha two tailed
Statistical Analysis 2: Comparison: Control (On Protocol Sample) vs Intervention (On Protocol); For the on protocol sample, study arm was associated with perfect ACTG-assessed 3-day ARV adherence at p = 0.024, alpha two-tailed; Test type: Superiority or Other; p = 0.024, HLM — The p-value was not adjusted for multiple comparisons, and thresholds for significance was 0.05 alpha, two tailed

2. Secondary Outcome: Viral Load Count
Description: Viral load data extracted from medical records beginning 30 days prior to baseline.
Time Frame: Measured over 18 months
Measure: Number; unit: percentage with undetectable viral load
Groups:
- Control (ITT Sample): 287 (94%) of the 304 randomized to control
Arm/Group | Control (ITT Sample) | Intervention (ITT Sample)
Number analyzed (Participants) | 287 | 277
percentage with undetectable viral load
  Baseline to 3 months (%) | 73.9 | 70.3
  3-6 months (%) | 70.3 | 77.0
  6-9 months (%) | 73.4 | 75.0
  9-12 months (%) | 76.1 | 76.8
  12-15 months (%) | 70.2 | 76.5
  15-18 months (%) | 74.5 | 79.3
Statistical Analysis 1: Comparison: Control (ITT Sample) vs Intervention (ITT Sample); For the ITT or OP samples, the significance threshold between groups over time for differential increases in proportion with suppressed (undetectable) viral load was p > 0.50. The study was underpowered to detect differences in Viral load; Test type: Superiority or Other; p > 0.50, Generalized Linear Model (GLM) — No adjustments were made

3. Primary Outcome: Visual Analog Scale Measure of Adherence to ART
Description: This measure asks participants to rate their adherence over the past 3 to 4 weeks using a line that marks from 0 to 100% of doses taken. For this study, this item was asked for each antiretroviral in one's regimen and a total score was produced by averaging all reports. For main outcomes, perfect vs imperfect adherence was evaluated.
  See: Walsh JC, Mandalia S, Gazzard BG. Responses to a 1 month self-report on adherence to antiretroviral therapy are consistent with electronic data and virological treatment outcome. AIDS.2002;16:269-77
Time Frame: Measured at each clinical visit over 18 months of participation
Population: Intent to treat included all participants with >=2 adherence assessments; OP sample further restricted this sample to those with >=6 assessments and no treatment interruptions over 18-months of participation. Multiple pairwise comparisons replaced missing values. HLM was used for over-time analyses on proportion reporting perfect adherence.
Measure: Number; unit: percent with 100% adherence
Groups:
- Intervention (On Protocol Sample): 152 (55%) of the ITT included intervention arm participants
Arm/Group | Control (ITT Sample) | Intervention (ITT Sample) | Control (On Protocol Sample) | Intervention (On Protocol Sample)
Number analyzed (Participants) | 287 | 277 | 176 | 152
percent with 100% adherence
  1 LifeWindows Visit (%) | 42.61 | 46.15 | 45.71 | 45.33
  2 LifeWindows Visits (%) | 43.27 | 47.81 | 43.35 | 47.37
  3 LifeWindows Visits (%) | 42.69 | 47.77 | 42.05 | 49.67
  4 LifeWindows Visits (%) | 42.21 | 48.44 | 40.34 | 44.74
  5 LifeWindows Visits (%) | 42.79 | 50.99 | 41.14 | 50.99
  6 LifeWindows Visits (%) | 45.83 | 49.12 | 45.98 | 51.32
  7 LifeWindows Visits (%) | 41.89 | 41.67 | 40.60 | 46.15
  8 LifeWindows Visits (%) | 35.09 | 40.63 | 34.00 | 42.35
  9 LifeWindows Visits (%) | 31.46 | 38.57 | 30.26 | 39.39
  10 LifeWindows Visits (%) | 29.41 | 36.84 | 28.07 | 36.54
  11 LifeWindows Visits (%) | 27.66 | 30.95 | 23.68 | 29.73
  12 LifeWindows Visits (%) | 28.13 | 31.25 | 23.08 | 23.08
  13 LifeWindows Visits (%) | 28.00 | 41.67 | 25.00 | 33.33
  14 LifeWindows Visits (%) | 23.08 | 42.86 | 10.00 | 27.27
Statistical Analysis 1: Comparison: Control (ITT Sample) vs Intervention (ITT Sample); For the ITT sample (t=586) the observed pattern of an increasing proportion of participants in the intervention arm reporting perfect adherence as time progressed from baseline was associated with a p-value of 0.12, alpha 0.05 two-tailed; Test type: Superiority or Other; p = 0.12, HLM — The p-value was not adjusted for multiple comparisons and is reported as 0.12 at alpha 0.05 two tailed
Statistical Analysis 2: Comparison: Control (On Protocol Sample) vs Intervention (On Protocol Sample); For the on protocol sample the pattern of increased proportion of participants in the intervention arm reporting perfect adherence as time progressed from baseline was associated with a p-value of 0.12, alpha 0.05 two-tailed; Test type: Superiority or Other; p = 0.12, HLM — The p-value was not adjusted for multiple comparisons, and is reported as 0.12 at alpha 0.05 two tailed

4. Post Hoc Outcome: Percentage of Participants Unemployed and on Disability
Time Frame: Data collected at Baseline
Measure: Number; unit: percentage of participant
Groups:
- On Protocol (OP) Sample: Post-hoc analysis of the participants provided >=6 assessments with no ART receipt interruptions
- Total Excluded From OP Sample: ITT sample excluded from the post-hoc analysis of the participants provided >=6 assessments with no ART receipt interruptions (ITT - OP sample)
Arm/Group | On Protocol (OP) Sample | Total Excluded From OP Sample
Number analyzed (Participants) | 328 | 266
percentage of participant
  % of participants Unemployed | 67 | 52
  % of participants on Disability | 55 | 43
Statistical Analysis 1: Comparison: On Protocol (OP) Sample vs Total Excluded From OP Sample; P-value for difference in unemployment rate between On Protocol (OP) sample, and participants excluded from on protocol analysis; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: On Protocol (OP) Sample vs Total Excluded From OP Sample; P-value for difference of participants on disability between On Protocol (OP) sample, and participants excluded from on protocol analysis; Test type: Superiority or Other; p < 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: Patient enrollment to end of IRB annual renewals
Description: No adverse events occurred during the study
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 0/304 | 0/290
Other Adverse Events (participants affected / at risk) | 0/304 | 0/290

LIMITATIONS AND CAVEATS:
* The only empirical demonstration of LifeWindows outcomes to date
* OP sample was defined a posteriori
* Under-powered to detect changes in Viral Load

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No